CLINICAL TRIAL: NCT00992225
Title: Phase 2 Evaluation of a Once Every 28 Days Dosing Regimen for LY573636-sodium in Patients With Metastatic Breast Cancer
Brief Title: A Study of LY573636-sodium in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12265; H8K-MC-JZAL (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: Metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY573636-sodium (Experimental)
  Interventions: Drug: LY573636-sodium

INTERVENTIONS:
Drug: LY573636-sodium — Dose is adjusted to target a specific maximum concentration (Cmax) based on patient laboratory parameters, administered intravenously every 28 days until disease progression or other criteria for patient discontinuation are met
  Other Names: tasisulam

SUMMARY:
The primary purpose of this study is to determine the objective response rate (complete and partial response) for patients who receive LY573636-sodium for metastatic breast cancer.

DETAILED DESCRIPTION:
Patient will receive a 2-hour intravenous infusion of study drug (LY573636-sodium) once every 28 days. Radiologic imaging scans will be performed before the first dose of study drug and then after every other treatment. Patients will be assessed for clinical progression at every visit and for response approximately every 56 days (every other cycle).

ELIGIBILITY:
Inclusion Criteria:

* Received at least 2 or more prior chemotherapy regimens for metastatic breast cancer.
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 4 weeks. Patients who have received whole-brain radiation must wait 90 days.

Exclusion Criteria:

* Serious pre-existing medical condition.
* Have active central nervous system or leptomeningeal metastasis.
* Current hematologic malignancies, acute or chronic leukemia.
* Receiving Warfarin (Coumadin).
* Have a history of radiation therapy involving more than 25% of the bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Temple, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- LY573636-sodium: Dose was adjusted to target a specific maximum concentration (Cmax) based on patient laboratory parameters, administered intravenously every 28 days until disease progression or other criteria for patient discontinuation were met
Period: Overall Study
Arm/Group | LY573636-sodium
Started | 43
Received at Least One Dose of Study Drug | 33
Completed | 33
Not Completed | 10
Not completed — Entry Criteria Not Met | 8
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | LY573636-sodium
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.43 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 3
  White | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  Participants
    0 - Fully active | 10
    1 - Ambulatory, restricted strenuous activity | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Overall Response
Description: Objective overall response is complete response (CR) + partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. It is calculated as a total number of participants with CR or PR divided by the total number of participants treated multiplied by 100.
Time Frame: Baseline to measured progressive disease or death from any cause up to 12 months
Population: All participants who received at least one dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | LY573636-sodium
Number analyzed (Participants) | 33
percentage of participants | 6.1 [1.1 to 17.9]

2. Secondary Outcome: Progression-free Survival
Description: Defined as the time from date of first dose to the first observation of progression of disease (PD) or death due to any cause. PD was determined using RECIST criteria. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Baseline to measured progressive disease or death from any cause up to 12 months
Population: All participants who received at least 1 dose of the study drug.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY573636-sodium
Number analyzed (Participants) | 33
months | 1.81 [1.64 to 2.17]

3. Secondary Outcome: Percentage of Participants Experiencing Clinical Benefit [(CR) + (PR) + Stable Disease (SD)]
Description: Clinical Benefit Rate = [(CR) + (PR) + Stable Disease (SD)] of at least 4 cycles/N as classified by the investigator according to the RECIST guidelines, where N = total number of participants with at least one dose of study drug. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: Baseline to measured progressive disease or death from any cause up to 12 months
Population: All participants who received at least one dose of the study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | LY573636-sodium
Number analyzed (Participants) | 33
percentage of participants | 9.1 [0.9 to 17.3]

4. Secondary Outcome: Duration of Overall Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. CR or PR is classified by the investigators according to RECIST guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions.
Time Frame: Time of response to progressive disease or death up to 12 months
Population: Zero participants analyzed. Duration of Overall Response for CR and PR data was not collected for analysis.
Arm/Group | LY573636-sodium
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Stable Disease
Description: Duration of stable disease (SD) is defined from date of documented SD to first date of progressive disease (PD) or death from any cause (assessed every other cycle during study therapy, or every 2 months during post-therapy). SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PR is ≥30% decrease in sum of longest diameter of target lesions. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Time from documented Stable Disease (SD) to first date of progressive disease or death from any cause up to 12 months
Population: All participants who received at least one dose of the study drug.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY573636-sodium
Number analyzed (Participants) | 33
months | 3.52 [3.45 to 3.98]

6. Secondary Outcome: The Percentage of Participants With Exposures in the Target Range
Description: Exposure is the amount of drug the body sees in a period of time. Target range is an exposure thought to offer the optimal balance of safety and efficacy based on prior research.
Time Frame: After drug infusion in cycles 1 and 2 (5 samples drawn over each 28 day cycle)
Population: All participants who received at least one dose of the study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | LY573636-sodium
Number analyzed (Participants) | 33
Percentage of participants
  Cycle 1 | 45
  Cycle 2: number analyzed (Participants) | 23
  Cycle 2 | 52

7. Secondary Outcome: Maximum Concentration (Cmax)
Time Frame: After drug infusion in cycles 1 and 2 (5 samples drawn over each 28 day cycle)]
Population: All participants who received at least one dose of the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Arm/Group | LY573636-sodium
Number analyzed (Participants) | 33
microgram/milliliter (µg/mL)
  Cycle 1 | 375 (16.4)
  Cycle 2: number analyzed (Participants) | 23
  Cycle 2 | 339 (17.2)

ADVERSE EVENTS:
Description: Adverse events (AEs) provided for all participants who received at least one dose of study drug. AEs are both study-drug related and non-study drug related. AEs represent all grades (1-5). Grade 1: mild adverse event (AE); Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening or disabling AE; Grade 5: death-related to AE.
Arm/Group | LY573636-sodium
Serious Adverse Events (participants affected / at risk) | 10/33
Other Adverse Events (participants affected / at risk) | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY573636-sodium (N=33)
Constipation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY573636-sodium (N=33)
Anaemia (Blood and lymphatic system disorders) | 5 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 11 (11)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (11)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (6)
Chest pain (General disorders) | 2 (2)
Fatigue (General disorders) | 21 (23)
Mucosal inflammation (General disorders) | 2 (3)
Oedema peripheral (General disorders) | 4 (4)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4)
Alanine aminotransferase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Blood alkaline phosphatase increased (Investigations) | 5 (5)
Blood creatinine increased (Investigations) | 2 (2)
Urine colour abnormal (Investigations) | 2 (2)
Weight decreased (Investigations) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 5 (5)
Renal failure (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days